CLINICAL TRIAL: NCT01150058
Title: Preclinical Evaluation of Novel CD33-Targeting Therapeutics for Treatment of Acute Myeloid Leukemia (AML)
Brief Title: Drug Biomarkers in Cell Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B19; COG-AAML10B19 (Other: Children's Oncology Group); NCI-2011-02241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML10B19 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-06-23; First posted 2010-06-24 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); childhood acute myeloid leukemia/other myeloid malignancies; adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — Blotting, Western; Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cell samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: western blotting
Other: flow cytometry
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying cell samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer

PURPOSE: This research study is studying drug biomarkers in cell samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine, in vitro, the cytotoxic activity of novel CD33-targeting immunoconjugate agents in cell samples from patients with acute myeloid leukemia (AML).
* To define the characteristics of AML cells responding to or resisting these agents.

OUTLINE: Cell samples are thawed and used for in vitro studies to determine the cytotoxic activity of novel CD33-targeting immunoconjugate agents, including gemtuzumab ozogamicin, for genotyping characterization by flow cytometry-based assays and/or western blot, and colony-forming cell assays.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia
* Cryopreserved samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients With Acute Myeloid Leukemia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Activity of novel CD33-targeting immunoconjugate agents
Genotypic characteristics of acute myeloid leukemia cells

CONTACTS AND LOCATIONS:
Overall Officials: Soheil Meshinchi, MD, Principal Investigator — Fred Hutchinson Cancer Center